CLINICAL TRIAL: NCT00215930
Title: Phase II Study on the Use of Molecular Analyses-Based Customized Chemotherapy in Patients With Stage IV/IIIB (Malignant Pleural Effusion) Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: The 'MADe IT' Clinical Trial: Molecular Analyses Directed Individualized Therapy for Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13208
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Results first posted 2011-02-23 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2011-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: malignant pleural effusion
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Pleural Effusion, Malignant | interventions — Vinorelbine; Docetaxel; Gemcitabine; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Double Agent Chemotherapy (Experimental): Molecular Analysis-Directed Chemotherapy Assignment based on gene expression of ERCC1 and RRM1.
  Interventions: Drug: Vinorelbine; Drug: Docetaxel; Drug: Gemcitabine; Drug: Carboplatin

INTERVENTIONS:
Drug: Vinorelbine — Ribonucleotide reductase subunit 1(RRM1)above 16.5 and Excision repair cross-complementing group 1 gene(ERCC1)above 8.7: Treat patients with Docetaxel and Vinorelbine (DV). DV group was treated with vinorelbine (45mg/m2ondays 1 and 15) and docetaxel (60mg/m2ondays 1 and 15) every 28 days.
  Other Names: Navelbine
Drug: Docetaxel — RRM1 below 16.5 and ERCC1 above 8.7: Treat patients with Gemcitabine and Docetaxel (GD). GD group was treated with gemcitabine (1,250 mg/m2 on days 1 and 8) and docetaxel (40 mg/m2 on days 1 and 8) every 21 days.
  RRM1 above 16.5 and ERCC1 below 8.7: Treat patients with Docetaxel and Carboplatin (DC). DC group was treated with docetaxel (75 mg/m2 on day 1) and carboplatin (AUC 5 on day 1) every 21 days.
  RRM1 above 16.5 and ERCC1 above 8.7: Treat patients with Docetaxel and Vinorelbine (DV). DV group was treated with vinorelbine (45mg/m2ondays 1 and 15) and docetaxel (60mg/m2ondays 1 and 15) every 28 days.
  Other Names: Taxotere
Drug: Gemcitabine — Ribonucleotide reductase subunit 1(RRM1) below 16.5, and Excision repair cross-complementing group 1 gene(ERCC1) below 8.7: Patients treated with Gemcitabine and Carboplatin (GC). GC group was treated with gemcitabine (1,250 mg/m2 on days 1 and 8) and carboplatin (area under the concentration-time curve [AUC] of 5 on day 1) every 21 days.
  RRM1 below 16.5 and ERCC1 above 8.7: Treat patients with Gemcitabine and Docetaxel (GD). GD group was treated with gemcitabine (1,250 mg/m2 on days 1 and 8) and docetaxel (40 mg/m2 on days 1 and 8) every 21 days.
  Other Names: Gemzar
Drug: Carboplatin — Ribonucleotide reductase subunit 1(RRM1) below 16.5, and Excision repair cross-complementing group 1 gene(ERCC1) below 8.7: Patients treated with Gemcitabine and Carboplatin (GC). GC group was treated with gemcitabine (1,250 mg/m2 on days 1 and 8) and carboplatin (area under the concentration-time curve [AUC] of 5 on day 1) every 21 days.
  RRM1 above 16.5 and ERCC1 below 8.7: Treat patients with Docetaxel and Carboplatin (DC). DC group was treated with docetaxel (75 mg/m2 on day 1) and carboplatin (AUC 5 on day 1) every 21 days.
  Other Names: Paraplatin

SUMMARY:
The standard treatment for non-small cell lung cancer, stage IV or IIIB malignant pleural effusion is chemotherapy. The decision to use a regimen is currently determined by toxicity or by physician's preference. In this protocol, the treatment regimen will be assigned based on the patients' tumor molecular profile. A tumor molecular profile analysis will allow the physician to define a specific molecular portrait that shows the genetic basis of the tumor. This analysis results in a detailed report that will determine which chemotherapy will be assigned to the patient.

DETAILED DESCRIPTION:
Evaluation at study entry will include blood tests, computerized tomography (CT) scans or other types of scans needed to measure other disease sites. A biopsy of one tumor is required for tumor analysis. If the patient's cancer has spread to other locations that may be easier to obtain tissue from and be less invasive, then the biopsy specimen may be collected from one of several possible locations that may exist within the patient's body. These possible sites include lung, bone, liver, adrenal glands, lymph nodes, nodules under the skin, or in cases of brain involvement requiring surgery, brain tissue. Sometimes fluids build up between the lining of the lung and the lung itself. If this happened to the patient and their doctor tells them the fluid should be drained, then this fluid may also be a source of cells we can use to analyze the patients cancer. In very rare cases, other sites might be identified.

Chemotherapy will consist of the assigned two drugs. Chemotherapy will be repeated every three or four weeks for at least two times. Patients will then have a CT scan to measure their tumor's response. Response can be reduction of tumor size, no change of tumor size, or increased tumor size. Doing CT Scans or other tests after every two cycles of chemotherapy will assess for response. If we see a favorable response we will continue chemotherapy for a maximum of two times after the best response we can see in the patient's tumor. If the patient's tumor grows larger, then we discontinue the study and the patient will discuss other treatment options with their doctor.

During treatment, a blood specimen will be obtained to check the patient's blood counts at the beginning and end of study, and prior to administration of every dose of chemotherapy. Approximately 3 teaspoonfuls (15 mls) of blood will be drawn each time.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed adenocarcinoma, large cell or squamous cell carcinoma NSCLC; as well as be willing to undergo a biopsy to enable customization of chemotherapy; unresectable/ metastatic (stage IV or IIIB malignant pleural effusion) NSCLC;
* male or female, aged > 18 years;
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1;
* adequate bone marrow, hepatic and renal function assessed within 14 days as evidenced by the following:

  1. absolute neutrophil count > 1,500/mm3
  2. platelet count > 100,000/mm3
  3. Hemoglobin > 8gm/dl
  4. no evidence of myelodysplastic syndrome or abnormal bone marrow reserve;
  5. creatinine < 1.5 x upper normal limit(UNL)
  6. total bilirubin must be within normal limits
  7. aspartate aminotransferase(AST)Serum glutamic oxaloacetic transaminase(SGOT) and/or alanine aminotranserase (ALT) serum glutamic pyruvic transaminase(SGPT) < 2×5 x UNL in the presence of a normal alkaline phosphatase;
  8. alkaline phosphatases < 4 x UNL in the presence of normal AST and ALT; patients with elevations of both alkaline phosphatase and liver enzymes (AST & ALT) will be excluded.
  9. serum calcium < 1.1 x UNL;
* at least one unidimensionally measurable lesion;
* signed informed consent;
* Women of childbearing potential should have negative pregnancy test prior to enrollment to study.
* Men with partners in the childbearing age group and women of childbearing potential must use effective contraception while on treatment and for 6 months thereafter.
* previous surgery (more that 30 days before study entry) is allowed but metastatic disease must be demonstrated;
* previous radiotherapy is allowed if:

  1. end of radiotherapy 21 days or more prior to study entry;
  2. patient has fully recovered from all toxic effects;
  3. at least one of the measurable target lesions is outside the radiation field.
* The patient will be enrolled and re-biopsied at the H Lee Moffitt Cancer Center. However since the patients are being treated by FDA approved drugs and with regimens for which phase I, phase II or phase III data are available the patients may have their chemotherapy administered at the their primary (referring) oncologists office.
* Complete initial staging work-up within 4 weeks prior to first infusion of chemotherapy.
* Patient should have a normal Prothrombin Time (PT) and Activated Prothrombin Time with Thromboplastin and kaolin (APTT), to enable him to undergo a biopsy.
* Peripheral neuropathy < grade I (according to the NCI-Common Terminology Criteria for Adverse Events (CTCAE Version 3.0)
* Patients with stable brain metastases will be allowed to enroll. Stable brain metastases being defined as no progression of brain metastases 28 days after conclusion of definitive treatment as documented by a CT Scan or MRI of the Brain

Exclusion Criteria:

* Pregnant or lactating women
* Prior systemic chemotherapy or immunotherapy for advanced NSCLC, patients may have received neoadjuvant or adjuvant therapy but more than 6 months prior to study entry;
* Prior malignancies, except cured non-melanoma skin cancer, curatively treated in situ carcinoma of the cervix or other cancer curatively treated and with non-evidence of disease for at least 3 years;
* presence of uncontrolled brain or leptomeningeal metastases;
* current peripheral neuropathy and hearing deficit of neural origin, CTCAE v3.0 grade 2 except if due to trauma;
* other serious illness or medical condition, including but not limited to:

  1. congestive heart disease; prior myocardial infarction within 6 months;
  2. history of significant neurologic or psychiatric disorders that would inhibit their understanding and giving of informed consent;
  3. infection requiring I.V. antibiotics and tuberculosis under treatment ongoing at study entry;
  4. untreated superior vena cava syndrome;
  5. active peptic ulcer; unstable diabetes mellitus or other contraindication to high dose corticosteroid therapy such as herpes, herpes zoster, cirrhosis;
  6. hypercalcemia requiring therapy at the time of study entry;
  7. preexisting clinically significant ascites and/or clinical significant pericardial effusion;
* patients whose lesion(s) are assessable only by radionuclide scan;
* patients with a history of severe hypersensitivity reaction to Taxotere or other drugs formulated with polysorbate 80 must be excluded
* concurrent treatment with other investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2004-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerold Bepler, MD, PhD, Principal Investigator — H. Lee Moffitt Cancer Center & Research Institute (now at Karmanos Cancer Institute)
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Assignments: High ERCC1 expression and High RRM1 Expression - vinorelbine plus docetaxel (DV); High ERCC1 expression but NOT High RRM1 expression - docetaxel plus gemcitabine (GD); High ERCC1 expression, but HAVE High RRM1 - carboplatin plus docetaxel (DC); High ERCC1 expression and do NOT have High RRM1 - carboplatin plus gemcitabine (GC)
Groups:
- Double Agent Chemotherapy: Molecular Analysis-Directed Chemotherapy Assignment based on gene expression of Ribonucleotide reductase subunit 1(ERCC1) and Excision repair cross-complementing group 1 gene (RRM1). GD group was treated with gemcitabine (1,250 mg/m2 on days 1 and 8) and docetaxel (40 mg/m2 on days 1 and 8) every 21 days. DC group was treated with docetaxel (75 mg/m2 on day 1) and carboplatin (AUC 5 on day 1) every 21 days. DV group was treated with vinorelbine (45mg/m2ondays 1 and 15) and docetaxel (60mg/m2ondays 1 and 15) every 28 days. GC group was treated with gemcitabine (1,250 mg/m2 on days 1 and 8) and carboplatin (area under the concentration-time curve [AUC] of 5 on day 1) every 21 days.
Period: Overall Study
Arm/Group | Double Agent Chemotherapy
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Double Agent Chemotherapy: Molecular Analysis-Directed Chemotherapy Assignment based on gene expression.
Arm/Group | Double Agent Chemotherapy
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 16
Age, Customized [Median (Full Range); unit: years] | 63 [38 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: Best Disease Response After a Maximum of Six Cycles.
Description: Determine the number of participants for each category of response rates (RR) in newly diagnosed patients with advanced non-small cell lung cancer (NSCLC) who are treated with a chemotherapeutic regimen assigned to them on the basis of expression of the genes ribonucleotide reductase subunit 1 (ERCC1) and excision repair cross-complementing group 1 gene (RRM1) expression. Prior to treatment we measured the level of ERCC1 and RRM1 expression in the patients tumor, on the basis of which the patient would be assigned a specific doublet chemotherapy.
Time Frame: 24 Months
Population: All participants were analyzed according to Response Evaluation Criteria in Solid Tumors (RECIST).
Measure: Number; unit: Participants
Groups:
- Double Agent Chemotherapy: Molecular Analysis-Directed Chemotherapy Assignment based on gene expression. Complete Response (CR): disappearance of all target lesions. Partial Response (PR): at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as reference the baseline sum LD. Progressive Disease (PD): at least a 20% increase in the sum of LD of target lesions taking as references the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD taking as references the smallest sum LD since the treatment started.
Arm/Group | Double Agent Chemotherapy
Number analyzed (Participants) | 53
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 23
  Stable Disease (SD) | 23
  Progressive Disease (PD) | 6
  Not Assessible | 1

2. Secondary Outcome: Overall Survival (OS)
Description: Median Overall Survival of Participants. OS and Progression Free Survival (PFS) probabilities were estimated using the Kaplan-Meier method. For statistical purposes, it is important to note that this trial was not designed to compare outcomes among patients assigned to the different chemotherapies, but rather that molecular analysis directed individualized chemotherapy assignment is feasible and yields promising results in outcomes.
Time Frame: 24 Months
Population: Review of all participants per protocol for Number at risk, Number of events, Number censored.
Measure: Median (Full Range); unit: Months
Arm/Group | Double Agent Chemotherapy
Number analyzed (Participants) | 53
Months | 13.3 [6 to 24]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was recorded as the time elapsed from the date of first treatment to the date of first evidence for disease progression or death. OS and PFS probabilities were estimated using the Kaplan-Meier method. For statistical purposes, it is important to note that this trial was not designed to compare outcomes among patients assigned to the different chemotherapies, but rather that molecular analysis directed individualized chemotherapy assignment is feasible and yields promising results in outcomes.
Time Frame: 24 Months
Population: Review of all participants for Number at risk, Number of events, Number censored.
Measure: Median (Full Range); unit: Months
Arm/Group | Double Agent Chemotherapy
Number analyzed (Participants) | 53
Months | 6.6 [6 to 24]

ADVERSE EVENTS:
Time Frame: 24 Months
Description: Toxicity was recorded according to the Common Terminology Criteria for Adverse Events version 3 (http://ctep.cancer.gov).
Arm/Group | Double Agent Chemotherapy
Serious Adverse Events (participants affected / at risk) | 29/53
Other Adverse Events (participants affected / at risk) | 5/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Agent Chemotherapy (N=53)
Allergic Reaction - Grade 3 (General disorders) | 1 (1) — Causality: Probably Related
Anemia - Grade 3 (Blood and lymphatic system disorders) | 1 (1) — Causality: Possibly Related
Cough - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Death not associated with CTCAE term - Grade 5 (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Probably Related
Dehydration - Grade 5 (General disorders) | 1 (1) — Causality: Possibly Related
Dyspnea - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Causality: 1 Probably Related, 1 Unknown
FN-ANC <1.0/Fever >=38.5C - Grade 3 (General disorders) | 2 (2) — Causality: 1 Possibly Related, 1 Unknown
Fatigue - Grade 3 (General disorders) | 4 (5) — Causality: 2 Probably Related, 1 Possibly Related, 2 Unknown
Hand/Foot Syndrome - Grade 3 (General disorders) | 2 (2) — Causality: 1 Probably Related, 1 Definitely Related
Hemoglobin - Grade 3 (Blood and lymphatic system disorders) | 2 (2) — Causality: Unknown
Hyperglycemia - Grade 3 (Blood and lymphatic system disorders) | 2 (2) — Causality: Unknown
Hypokalemia - Grade 3 (Blood and lymphatic system disorders) | 2 (2) — Causality: Unknown
Hyponatremia - Grade 3 (General disorders) | 3 (4) — Causality: Unknown
Hypoxia - Grade 3 (General disorders) | 1 (1) — Causality: Probably Related
International Normalization Ratio (INR) - Grade 3 (General disorders) | 1 (1) — Causality: Unknown
Intracranial Hemorrhage - Grade 5 (Vascular disorders) | 1 (1) — Causality: Probably Related
Lacrimation - Grade 3 (General disorders) | 1 (1) — Causality: Probably Related
Leukocytes - Grade 3 (Blood and lymphatic system disorders) | 7 (9) — Causality: 1 Probably Related, 4 Unknown
Lymphocytes - Grade 3 (Blood and lymphatic system disorders) | 11 (11) — Causality: Unknown
Nail Changes - Grade 3 (General disorders) | 1 (1) — Causality: Definitely Related
Neuropathy-Motor - Grade 3 (General disorders) | 1 (1) — Causality: Possibly Related
Neuropathy-Sensory - Grade 3 (General disorders) | 1 (1) — Causality: Possibly Related
Neutropenia - Grade 3 (General disorders) | 2 (3) — Causality: Probably Related
Neutropenia - Grade 4 (General disorders) | 1 (1) — Causality: Probably Related
Neutrophils - Grade 3 (General disorders) | 5 (5) — Causality: Unknown
Pain/Nausea/Vomiting - Grade 3 (General disorders) | 1 (1) — Causality: Probably Related
Pedal Edema - Grade 3 (General disorders) | 1 (1) — Causality: Probably Related
Platelet Count - Grade 3 (Blood and lymphatic system disorders) | 1 (1) — Causality: Unknown
Pulmonary Embolism - Grade 4 (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Not Related
RLL DVT - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Causality: Possibly Related
Syncope - Grade 3 (Vascular disorders) | 1 (1) — Causality: Possibly Related
Thrombocytopenia - Grade 3 (Blood and lymphatic system disorders) | 1 (1) — Causality: Probably Related
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Agent Chemotherapy (N=53)
Hemoglobin - Grade 1 (Blood and lymphatic system disorders) | 1 (1) — Causality: Unknown
Hypokalemia - Grade 1 (Blood and lymphatic system disorders) | 1 (1) — Causality: Unknown
Leukocytes - Grade 1 (Blood and lymphatic system disorders) | 1 (2) — Causality: Unknown
Lymphocytes - Grade 1 (Blood and lymphatic system disorders) | 1 (1) — Causality: Unknown
Platelet Count - Grade 1 (Blood and lymphatic system disorders) | 1 (1) — Causality: Unknown

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No